CLINICAL TRIAL: NCT04708158
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Aerosolized Novaferon vs. Placebo in Hospitalized Adult Patients With ModerateCOVID-19
Brief Title: Novaferon for COVID-19 Treatment Trial (NCTT-005)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genova Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JH-COR-005
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: antiviral; SARS-CoV-2; COVID19
MeSH Terms: conditions — COVID-19 | interventions — recombinant interferon alpha 2b-like protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Inhaled Novaferon, given 20 ug BID, daily for 7 days
  Interventions: Biological: Novaferon
- Placebo (Placebo Comparator): Inhaled saline (placebo), given BID, daily for 7 days
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Novaferon — a novel recombinant antiviral protein drug
  Arms: Active
Biological: Placebo — Saline
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled trial for hospitalized moderate COVID-19 patients

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained from the participants with age of over 20 years at the time of signing the informed consent.
* SARS-CoV-2 infection is diagnosed by the positive SARS-CoV-2 detection of RT-PCR tests within 72 hours before the start of administration of the investigational drug
* Less than 6 days from onset of COVID-19 symptoms to starting the administration of the investigational drug. The symptoms are defined as one or more of the following: fever (37.5 ºC or higher), respiratory symptoms (cough, shortness of breath, chest pain, sore throat, running nose, nasal congestion, etc.), headache, malaise, abdominal pain, diarrhea, nausea, vomiting, loss of smell, loss of taste, or other COVID-19 symptoms defined by investigators or physicians.
* Have at least one of the following findings.
* Oxygen saturation (SpO2) measured by pulse oximeter is less than 96% and more than 93%.
* Chest X-ray or CT scan shows pneumonia findings suggestive of COVID-19 infection
* Need hospitalization and COVID-19-related medical care.
* Require no supplemental oxygen.
* Women (less than 12 months after the last menstrual period) who have a negative pregnancy test (urine hCG qualification) and agree to take oral contraceptives or use condom during study period.

Exclusion Criteria:

* History of hypersensitivity to interferon or Novaferon or any excipients of interferon or Novaferon.
* Having received other antiviral treatments (Favipiravir, Remdesivir, Interferon, etc.).
* CTCAE Grade 3 or higher liver dysfunction (ALT / AST> 5ULN) or renal dysfunction (eGFR <30 mL / min / 1.73 m2).
* Active infections or other medical conditions that contraindicate inhalation therapy.
* Inappropriate for inclusion in the clinical trial as determined by investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | From enrollment up to Day 28
  Time to patient clinical improvement by 2 points on a 7-point ordinal scale

SECONDARY OUTCOMES:
Rate of clinical improvement | Day 1 to Day 10, 14 and 28
  Rate at which patients show a clinical improvement by 2 points on a 7-point ordinal scale
Rate of clinical deterioration | Day 1 to Day 10, 14 and 28
  Rate at which patients show a clinical deterioration by 2 points on a 7-point ordinal scale
Time to viral clearance | From enrollment up to Day 28
  Time taken for patients to demonstrate negative RT-PCR test of SARS-CoV-2 in the samples taken from nasopharyngeal swabs
Rate of viral clearance | Each Day from Day 1 up to Day 28
  The rate at which patients demonstrate negative RT-PCR test of SARS-CoV-2 in the samples taken from nasopharyngeal swabs
Change in viral load | Each Day from Day 1 up to Day 28
  Changes of SARS-CoV-2 viral loads in the samples of nasopharyngeal swabs
Mortality rate | At Day 28
  Mortality rate
Duration of hospital stay | From enrollment up to Day 28
  Number of days the patient is in hospital
Time to resolution of symptoms | From enrollment up to Day 28
  Time taken for patients to demonstrate a resolution of symptoms defined as a (National Early Warning Score 2) NEWS 2 of 0 maintained for 24hours
Requirement of supplemental oxygen | From enrollment up to Day 28
  Rate at which patients require supplemental oxygen
Requirement of mechanical ventilation | From enrollment up to Day 28
  Rate at which patients require mechanical ventilation (invasive or non-invasive)
Rate of alive patients | At Day 28
  Rate of patients alive without having to use invasive ventilator or ECMO
Adverse events | From enrollment up to Day 28
  Adverse event incidence, type and severity

CONTACTS AND LOCATIONS:
Locations (22):
- Japan (22):
  - Chiba Aoba Municipal Hospital, Chiba
  - Kamagaya General Hospital, Chiba
  - NHO Chiba Medical Center, Chiba
  - NHO Omuta National Hospital, Fukuoka
  - NHO Kasumigaura Medical Center, Ibaraki
  - Tsukuba Medical Center Foundation Tsukuba Medical Center Hospital, Ibaraki
  - Kokankai Nippon Kokan Hospital, Kanagawa
  - Rakuwakai Otowa Hospital, Kyoto
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - Osaka Habikino Medical Center, Osaka
  - Rinku General Medical Center, Osaka
  - Sakai City Medical Center, Osaka
  - Omi Medical Center, Shiga
  - NHO Utsunomiya Hospital, Tochigi
  - Japanese Red Cross Medical Center, Tokyo
  - Juntendo University Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Showa University East Hospital, Tokyo
  - Showa University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - Tokyo Shinagawa Hospital, Tokyo
  - NHO Iwakuni Clinical Center, Yamaguchi